CLINICAL TRIAL: NCT02459184
Title: IGNITE (addressInG iNcome securITy in Primary carE) Study: A Pragmatic Randomized Controlled Trial
Brief Title: addressInG iNcome securITy in Primary carE
Acronym: IGNITE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SMH2015
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Poverty; Income; Social Determinants of Health
Keywords: preventive medicine; social determinants of health; primary health care; poverty; income; health promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention (Experimental): Participants will meet with the Income Security Health Promoter immediately.
  Interventions: Other: Income Security Health Promotion
- Late intervention (Active Comparator): Participants will meet with the Income Security Health Promoter at 6 months.
  Interventions: Other: Income Security Health Promotion

INTERVENTIONS:
Other: Income Security Health Promotion — The ISHP will work to improve the income security of participants within this study. To that end, her activities include:
  * Providing one-to-one case management support and ongoing follow-up to diverse low-income patients and families regarding their income security.
  * Developing and implementing targeted information self-help sessions, such as; banking basics, income tax submissions, and social service forms, for the target population
  * Developing and maintaining up-to-date detailed knowledge of financial issues and financial services affecting low-income people, and applying this knowledge in his/her work.
  * Assisting individual low-income patients with income security-focused interventions, including access to tax benefits, applications for income security programs such as social assistance and seniors and child benefits, and navigation of disability support programs.

SUMMARY:
Social processes that impact the health of individuals have been labeled the social determinants of health (SDOH). These are "the conditions in which people are born, grow, live, work and age. These circumstances are shaped by the distribution of money, power and resources at global, national and local levels". Perhaps the most important SDOH is income security, a person's actual, perceived and expected income. Our objective is to carry out a pragmatic randomized controlled trial that evaluates the impact of an income-focused health promoter.

DETAILED DESCRIPTION:
This study aims to answer the question: What is the impact of an income security health promotion service based in a primary care setting on the income security of people living in poverty? We hypothesize that an income security health promotion service for adults living in poverty will increase monthly income relative to usual care. We will carry out a pragmatic randomized controlled trial that evaluates the impact of such a new service focused on income security health promotion. The St. Michael's Hospital Academic Family Health Team has received ongoing funding from the Ministry of Health and Long-Term Care (MOHLTC) to support this service. The primary outcome is income security, and secondary outcomes include quality of life, financial literacy and community integration.

Population - Adults living in poverty Intervention - Income security health promotion Control - Usual care Outcome - Primary: Improvement in income per month in the intervention group at 6 months (post-intervention) compared to income in control group at 6 months (pre-intervention). Secondary: quality of life, self-rated health, community engagement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Lives within the Metropolitan catchment areas
* Lives in a postal code that is in the lowest income quintile, or has had a billing code specific to social assistance forms billed ever billed, or has been identified as low income based on reported family income and number of people supported by income on the "Health Equity Data"
* Patient of the Family Health team including those that are: rostered, non-rostered, refugee claimants (IFH) or uninsured seen in the FHT.
* Verified by the patient's family physician as living in poverty, a good candidate for the intervention, and the patient's family physician agrees to have a letter submitted with his/her name attached.

Exclusion Criteria:

* Patients who have previously worked with the Income Security Health Promoter, or are part of households of people who have previously worked with the Income Security Health Promoter.
* Patients who have no available contact information for mailing.
* Patients of any member of the investigative team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in monthly income from baseline to 6 months after intervention | 6 months
  Change in monthly income from baseline to 6 months after intervention

SECONDARY OUTCOMES:
quality of life: Change in scores on the WHO QoL-BREF and EQ-5D-5L | 12 months
  Change in scores on the WHO QoL-BREF and EQ-5D-5L
quality of life (overall health, mental health, physical health): change in units on a measured scale of EQ VAS | 12 months
  changes in units on a measured scale
community integration: Change in scores on the Community Integration Scale | 12 months
  Change in scores on the Community Integration Scale
financial literacy: Change in scores on the Canadian Centre for Financial Literacy Personal Financial Literacy Quiz | 12 months
  Change in scores on the Canadian Centre for Financial Literacy Personal Financial Literacy Quiz
co-morbidities and medication access | 12 months
  changes to scores relating to comorbidities and medication access
other social determinants | 12 months
  changes scores relating to housing and employment
food security | 12 months
  changes in scores on Health Canada food security module

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pinto, MD MSc, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
In consultation with our institutional Research Ethics Board, we will consider release of IPD to other researchers.